CLINICAL TRIAL: NCT00081588
Title: An Open Label Trial of TMC114/RTV in HIV-1 Infected, Treatment-experienced Subjects.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR006724; TMC114-C215; NCT00980226 (obsolete NCT alias)
Record Dates: First submitted 2004-04-15; First posted 2004-04-19 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: HIV Infection
Keywords: TMC114-C215; Ritonavir; HIV infections; TMC114-C202; TMC114-C213
MeSH Terms: conditions — HIV Infections | interventions — Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 001 (Experimental): TMC114600/100 mg tablets of TMC114/rtv BID for 144 weeks or until commercial available
  Interventions: Drug: TMC114

INTERVENTIONS:
Drug: TMC114 — 600/100 mg tablets of TMC114/rtv BID for 144 weeks or until commercial available

SUMMARY:
The primary objective of the TMC114-C215 study is to evaluate the safety and tolerability of TMC114/RTV over time. The secondary objectives are to evaluate the antiviral activity over time and to evaluate the immunological effect over time.

DETAILED DESCRIPTION:
The study will continue for 144 weeks after study medication has begun. For patients failing treatment, they must have participated in the TMC114-C213 or TMC114-C202 for at least 12 weeks and meet specific virologic failure criteria. It is estimated that approximately 150 patients may meet these criteria. Major inclusion and exclusion criteria are listed below. For new patients, they must have been on prior antiretroviral therapy, including more than one nucleoside reverse transcriptase inhibitor (NRTI), one non-nucleoside reverse transcriptase inhibitor (NNRTI) and a protease inhibitor (PI). At least one primary PI mutation must be present at screening. Many of the same centers that are participating in the TMC114-C213 and TMC-114 -C202 studies are also participating in the TMC114-C215 study. All sites have the chance to recruit rollover patients into the TMC114-C215 study and some sites listed had approval to recruit new patients into the study. The recruitment of new patients for the TMC114-C215 trial has been fully enrolled. The TMC114-C202 and TMC114-C213 have completed so no more patients are enrolled in this study. Two 300mg/100mg Darunavir/Ritonavir tablets twice daily for 144 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in the TMC114-C202 or TMC114-C213 trials
* Significant virologic failure during participation in the above trials
* Study participation in the treatment phase of the original trial for a total of at least 12 weeks before TMC114-C215 screening
* Patient agrees to take TMC114/RTV with at least 2 other antiretrovirals (NRTIs), with or without T-20, from baseline onwards
* Patient has given informed consent

Exclusion Criteria:

* Use of disallowed concomitant therapy
* Patient with clinical or laboratory evidence of active liver disease, liver impairment/ dysfunction or cirrhosis irrespective of liver enzyme levels
* Any active or unstable medical condition that, in the investigator's opinion, would compromise the subject's safety
* Patient with laboratory abnormalities at screening as defined by ACTG grading scheme as listed in the protocol
* Patient withdrawing consent from TMC114-C202 or TMC114-C213

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2003-11; Primary Completion 2005-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary parameter is the confirmed virologic response at Week 24 (a drop in viral load (copies/mL) of at least 1 log10 versus baseline. | 24 weeks

SECONDARY OUTCOMES:
Proportion of patients with a virologic response; with plasma HIV-1 RNA levels < 50 copies/mL; with plasma HIV-1 RNA levels < 400 copies/mL; Time to loss of virologic response over 144 week treatment period; Change in plasma viral load at all time points | 144 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited
Locations (64):
- United States (26):
  - Birmingham, Alabama
  - Beverly Hills, California
  - La Jolla, California
  - Long Beach, California
  - Los Angeles, California
  - Oakland, California
  - San Francisco, California
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Miami, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Macon, Georgia
  - Chicago, Illinois
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Camden, New Jersey
  - Albany, New York
  - New York, New York
  - Cincinnati, Ohio
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - Galveston, Texas
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Buenos Aires, Argentina
- Australia (3):
  - Darlinghurst
  - Melbourne
  - Perth
- Vienna, Austria
- Belgium (2):
  - Brussels
  - Ghent
- Brazil (4):
  - Campinas
  - Curitiba
  - Rio de Janeiro
  - São Paulo
- Canada (3):
  - Calgary, Alberta
  - Toronto, Ontario
  - Montreal, Quebec
- France (6):
  - Le Kremlin-Bicêtre
  - Montpellier
  - Nantes
  - Paris
  - Toulon
  - Villejuif
- Germany (9):
  - Berlin
  - Bonn
  - Düsseldorf
  - Essen
  - Freiburg im Breisgau
  - Hamburg
  - Kÿln
  - Mannheim
  - Munich
- Budapest, Hungary
- Portugal (2):
  - Lisbon
  - Porto
- Spain (3):
  - Barakaldo Vizcaya S/N
  - Barcelona
  - Madrid
- United Kingdom (3):
  - Edinburgh
  - London
  - Manchester

REFERENCES:
- [Result] Molina JM, Cohen C, Katlama C, Grinsztejn B, Timerman A, Pedro Rde J, Vangeneugden T, Miralles D, Meyer SD, Parys W, Lefebvre E; TMC114-C208 Study Group; TMC114-C215 Study Group. Safety and efficacy of darunavir (TMC114) with low-dose ritonavir in treatment-experienced patients: 24-week results of POWER 3. J Acquir Immune Defic Syndr. 2007 Sep 1;46(1):24-31. doi: 10.1097/QAI.0b013e3181359cfb. PMID 17621237